CLINICAL TRIAL: NCT07095140
Title: Assessing Co-Use of Oral Nicotine Pouches and Alcohol Among Young Adults
Brief Title: Studying the Effects of Nicotine Concentration and Flavor on Alcohol Use in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Brittney Keller-Hamilton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: OSU-24392; NCI-2025-04731 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Alcohol-Related Carcinoma
MeSH Terms: interventions — Ecological Momentary Assessment

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single blind study, meaning all participants will be blinded to the study product they use during each 10 day sampling period to avoid potential study bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low concentration, smooth-flavored (Experimental): Participant tries low concentration, Smooth-flavored oral nicotine pouches over a 10-day period in the absence of unacceptable toxicity. Participants also complete pre-scheduled EMAs over 10 minutes BID and as needed on the mornings after a drinking event during each 10-day ONP use period. Additionally, participants wear an alcohol monitoring wristband for at least 22 hours per day on study.
  Interventions: Other: Ecological Momentary Assessment; Other: Monitoring; Drug: Nicotine Oral Pouch; Other: Survey Administration
- High concentration, smooth-flavored (Experimental): Participant tries high concentration Smooth-flavored oral nicotine pouches over a 10-day period in the absence of unacceptable toxicity. Participants also complete pre-scheduled EMAs over 10 minutes BID and as needed on the mornings after a drinking event during each 10-day ONP use period. Additionally, participants wear an alcohol monitoring wristband for at least 22 hours per day on study.
  Interventions: Other: Ecological Momentary Assessment; Other: Monitoring; Drug: Nicotine Oral Pouch; Other: Survey Administration
- Low concentration, spearmint-flavored (Experimental): Participant tries low concentration spearmint-flavored oral nicotine pouches over a 10-day period in the absence of unacceptable toxicity. Participants also complete pre-scheduled EMAs over 10 minutes BID and as needed on the mornings after a drinking event during each 10-day ONP use period. Additionally, participants wear an alcohol monitoring wristband for at least 22 hours per day on study.
  Interventions: Other: Ecological Momentary Assessment; Other: Monitoring; Drug: Nicotine Oral Pouch; Other: Survey Administration
- High concentration, spearmint-flavored (Experimental): Participant tries high concentration spearmint-flavored oral nicotine pouches over a 10-day period in the absence of unacceptable toxicity. Participants also complete pre-scheduled EMAs over 10 minutes BID and as needed on the mornings after a drinking event during each 10-day ONP use period. Additionally, participants wear an alcohol monitoring wristband for at least 22 hours per day on study.
  Interventions: Other: Ecological Momentary Assessment; Other: Monitoring; Drug: Nicotine Oral Pouch; Other: Survey Administration

INTERVENTIONS:
Other: Ecological Momentary Assessment — Complete EMAs
  Other Names: EMA
Other: Monitoring — Wear alcohol monitoring wristband
  Other Names: monitor
Drug: Nicotine Oral Pouch — Receive ONPs
  Other Names: ZYN
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies the use of both (co-use) oral nicotine pouches (ONPs) and alcohol among young adults and whether ONP nicotine concentration and flavor affect alcohol use. The co-use of nicotine and alcohol has grown among young adults and the increase in ONP use among young adults may be a contributing factor. ONPs do not contain tobacco leaf and may reduce cancer risk for those who switch from traditional tobacco products (e.g., cigarettes, moist snuff) to ONPs. However, given that alcohol is a cancer-causing agent, using ONPs might increase alcohol use among young adults, which may cause an increase in their risk of cancer. ONPs come in different nicotine concentrations and flavors, with young adults expressing a preference in nicotine concentration or flavor for use while drinking. The different nicotine concentrations and flavors could lead users to drink more or longer. Studying the co-use of ONPs and alcohol among young adults may help researchers understand whether ONP nicotine concentrations and flavors affect alcohol use. This information may be used to help guide future ONP regulations and cancer prevention interventions targeted to young adults.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the role of ONP nicotine concentration on alcohol consumption and side effects during a drinking event.

II. Evaluate the role of ONP flavor on alcohol consumption and side effects of co-use during a drinking event.

III. Describe the effects of ONP nicotine concentration and flavors on next-day side effects after drinking events.

OUTLINE: Participants are randomized to a sequence of 4 ONP with different nicotine concentrations and flavors.

Participants receive four different types of ONPs consisting of low nicotine concentration, high nicotine concentration, unflavored, and spearmint on study. Participants then use the ONPs over 10 days in the order of the assigned sequence for a total of four 10-day periods in the absence of unacceptable toxicity. Participants also complete pre-scheduled ecological momentary assessments (EMAs) over 10 minutes twice daily (BID) and as needed on the mornings after a drinking event during each 10-day ONP use period. Additionally, participants wear an alcohol monitoring wristband for at least 22 hours per day on study.

ELIGIBILITY:
Inclusion Criteria:

* 21-30 years old
* Use ONPs daily
* Drink alcohol at least three days/week
* Read and speak English
* Own an iPhone (required for BACtrack Skyn wristband)
* Used 6 mg nicotine concentration ONPs on at least 20 days of past month

Exclusion Criteria:

* Use of other tobacco products > 10 days/month
* Unstable or significant medical condition
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* History of cardiac event or distress within the past three months
* Currently pregnant, planning to become pregnant within six months, or breastfeeding (all participants assigned female at birth will take a pregnancy test at each clinic visit before provision of study products; a negative test will be needed to proceed with product sampling)

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | Four 10-day ONP use periods
  Alcohol consumption will be estimated with transdermal alcohol content (TAC) collected with a wristband worn by the participants.
Alcohol and ONP co-use side effects | Four 10-day ONP use periods
  The incidence of side effects including nausea, dizziness, and "head buzz" will be evaluated with the EMA surveys administered on the days of alcohol and ONP co-use.
Alcohol and ONP co-use next-day side effects | Four 10-day ONP use periods
  The incidence of next-day side effects including nausea, fatigue, sleep disruptions, and shakiness will be evaluated with the EMA surveys administered on the morning after a day where alcohol and ONP were co-used.

CONTACTS AND LOCATIONS:
Overall Officials: Brittney L Keller-Hamilton, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu